CLINICAL TRIAL: NCT06993636
Title: Population Pharmacokinetic/Pharmacodynamic Analysis of Rivaroxaban in Chinese Children Aged Over 2 Years With Giant Coronary Artery Aneurysm After Kawasaki Disease
Brief Title: Pharmacometrics Analysis of Rivaroxaban in Chinese Children Aged Over 2 Years
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: RIVA-KD-PopPK
Record Dates: First submitted 2025-05-11; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Kawasaki Disease; Coronary Artery Aneurysm; Rivaroxaban; Anticoagulant Drugs; Pharmacokinetics and Pharmacodynamics
Keywords: Kawasaki disease; Coronary artery aneurysm; Population pharmacokinetic and pharmacodynamic; rivaroxaban; anticoagulant
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Coronary Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rivaroxaban: Rivaroxaban as anticoagulant will be administered with antiplatelet drug for long-term antithrombotic treatment, following a model-based optimized dosing regimen. Rivaroxaban plasma concentration and rivaroxaban-calibrated Anti-FXa activity are measured for clinical monitoring

SUMMARY:
Based on an established Kawasaki disease cohort database, this prospective, single-center, single-arm, observational study will collect clinical data from children aged 2 years and older with giant coronary artery aneurysms after Kawasaki disease who received rivaroxaban treatment. Rivaroxaban plasma concentrations, anti-factor Xa activity levels, and genetic polymorphisms will be measured and analyzed to support the population pharmacokinetic/pharmacodynamic analysis

ELIGIBILITY:
Inclusion Criteria:

1. Giant coronary artery aneurysm(s) in any coronary artery after acute stage of Kawasaki disease. Giant coronary artery aneurysm(s) should be confirmed by two-dimensional echocardiography and meet the diagnostic criteria of Z-score ≥10 or coronary artery internal diameter ≥8mm;
2. Anticoagulant with antiplatelet drug therapy for anti-thromboprophylaxis is recommended for the next 6 months;
3. Children aged 2 years to <18 years

Exclusion Criteria:

1. Active bleeding or bleeding risk contraindicating anticoagulant therapy
2. Hypersensitivity or any other contraindications listed in the local labeling for the comparator treatment or experimental treatment
3. Patients participating in clinical trials of other drugs at the same time

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged ≥2 years with giant coronary artery aneurysms after Kawasaki disease treated with rivaroxaban at the Children's Hospital of Fudan University
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rivaroxaban plasma concentration | From baseline to 6 months after rivaroxaban initiation, with scheduled sampling at the first hospitalization
  Opportunistic blood sampling will be performed at multiple predefined time points based on the principle of sparse sampling. It includes: 1. Day 1, 20 minutes -1 h after the first dose; 2. Day 1, 7±1 h after the first dose; 3. After at least three continuous doses (≥ Day 4): before the scheduled dose at that day, which is defined as the trough concentration; 4. After at least three continuous doses (≥ Day 4): 3±1 h the scheduled dose at that day, which is defined as the peak concentration. And peak and trough concentrations will be re-measured after each dose adjustment
Rivaroxaban-calibrated anti-activated Factor X (FXa) activity | From baseline to 6 months after rivaroxaban initiation, with anti-FXa activity measured at the same time points as plasma concentration
  Opportunistic blood sampling will be performed at multiple predefined time points based on the principle of sparse sampling. It includes: 1. Day 1, 20 minutes -1 h after the first dose; 2. Day 1, 7±1 h after the first dose; 3. After at least three continuous doses (≥ Day 4): before the scheduled dose at that day, which is defined as the trough concentration; 4. After at least three continuous doses (≥ Day 4): 3±1 h the scheduled dose at that day, which is defined as the peak concentration. And peak and trough concentrations will be re-measured after each dose adjustment

SECONDARY OUTCOMES:
Occurrence of new thrombosis in coronary arteries | From baseline to 6 months after rivaroxaban initiation
  It is binary variable. Every echocardiography conducted during study period will be documented. Researcher will document whether new thrombosis occurs in coronary arteries, and record the number of involved coronary arteries.
Composite of Major bleeding or Clinically relevant non-major bleeding event | From baseline to 6 months after rivaroxaban initiation
  It is a binary variable. Researcher will document major bleeding or clinically relevant non-major bleeding events. Major bleeding is defined as 1.Fatal bleeding; 2.Clinically overt bleeding associated with a decrease in Hemoglobin of ≥20 g/L in a 24-h period; 3.Critical site bleeding, such as retroperitoneal, pulmonary, pericardial, intracranial, or otherwise involves the central nervous system; 4.Bleeding that requires an intervention via an invasive procedure; 5.Overt bleeding for which a reversal agent is administered. Clinically relevant non-major bleeding event is defined as 1.Bleeding that results in a medical or procedural intervention not meeting major bleeding criteria, including a medication change (reducing, holding, or changing anticoagulation or addition of new medication) ; 2.Bleeding that results in hospitalization or increased level of care; 3.Overt bleeding for which a blood product is administered, and does not meet the criteria for major bleeding

OTHER OUTCOMES:
Genetic polymorphism | Day 1
  Opportunistic sampling will be performed using the remaining blood specimens collected for rivaroxaban plasma concentration measurement. Genetic polymorphisms related to rivaroxaban metabolism and transport will be examined, including CYP3A4, ABCB1, ABCG2, and et.cl CYP3A4: Cytochrome P450 Family 3 Subfamily A Member 4, ABCB1: ATP Binding Cassette Subfamily B Member 1; ABCG2: ATP Binding Cassette Subfamily G Member 2

CONTACTS AND LOCATIONS:
Overall Officials: Fang Liu, MD, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No